CLINICAL TRIAL: NCT05358366
Title: Infección de Amor (Love Infection): Online Delivery and Pilot Testing of a Dramatized Story Intervention (Telenovela/Soap Opera) for HIV Prevention Among Latinas in North Carolina
Brief Title: Love Infection: A Dramatized Story Intervention (Telenovela/Soap Opera) for HIV Prevention
Acronym: IA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-3214; 550KR262124 (Other Grant/Funding Number: NC TraCS NIH Clinical and Translational Science Award (CTSA))
Record Dates: First submitted 2022-04-26; First posted 2022-05-03 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-03

CONDITIONS: HIV Infections
Keywords: HIV; Latinas; Primary Disease Prevention; Internet Based Intervention
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: 2 arms, intervention and wait-listed control group. Participants in the intervention group will receive the 4 episodes of the Love infection intervention (one episode weekly) after the baseline assessment. Participants in the wait-listed control group will receive the intervention after completing the 3-month assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infeccion de Amor (Love Infection) (Experimental): 33 Latinas will view four IA intervention episodes, one per week immediately after the baseline survey and orientation.
  Participants will receive an email to their preferred email address with a password to access to the episode on the IA's website: https://www.infecciondeamor.com. Each 10-minute episode can be watched more than once during the week and presents a situation with notable HIV risk and ways the characters avoided risk (e.g., condom use) or confronted consequences of poor practices (e.g., HIV infection). The one-week time frame for each episode is needed to provide time to review and reflect about IA's content and modify HIV prevention behaviors. It will also allow Latinas to obtain information and support from the team and referral if needed. This time frame was effective to improve behaviors in previous studies.
  Interventions: Behavioral: Infeccion de Amor (Love Infection)
- Wait-listed (Other): A wait-listed control group of 33 Latinas will receive IA in the same manner as the intervention group.
  Latinas will start watching the telenovela episodes 4 months after their baseline survey (after T3 survey).
  Latinas will be informed at recruitment of this group condition and the study randomization. During the waiting time, participants will be called on a monthly basis to encourage participation and refer to services if needed.
  Interventions: Behavioral: Infeccion de Amor (Love Infection)

INTERVENTIONS:
Behavioral: Infeccion de Amor (Love Infection) — Love Infection is a filmed dramatized story (telenovela/soap opera) Infección de Amor (IA), or "Love Infection" - culturally tailored for US Latinas and delivered online. IA is a four-episode HIV prevention telenovela co-created with Latinas and a community-based participatory and interdisciplinary. Participants have one week window to watch the 10-minute episodes from their preferred device and location.

SUMMARY:
Purpose: To test the feasibility, acceptability of the IA intervention (four telenovela episodes), assessment of the mechanisms of action (self-efficacy, narrative engagement, and emotional elicitation) and conduct a randomized controlled pilot study to examine the change in primary outcomes (condom use, HIV testing, Pre-exposure Prophylaxis (PrEP) awareness and use) and secondary outcomes (Substance abuse (SA), intimate partner violence (IPV), and depression comparing 33 intervention- and 33 control Latinas at baseline (T1, pre-intervention), T2 (immediately post-intervention, 1 month) and T3 (3 months after the end of the intervention, with no intervening contact with study staff).

Participants: 66 Latinas ages 18-44 years who report sexual activity with a man in the last 6 months, have internet access from any device, and reside in NC.

Procedures (methods): Participants will be asked to: (1) receive an orientation about the use of the Infección de Amor (IA) telenovela website and access the telenovela website once a week for 4 weeks to watch a telenovela episode and answer some questions about the episode (half hour each week, 2 in total), (2) attend to a one hour-meeting with the research team to complete a baseline survey, (3) complete a survey (on their own) one-month after the baseline survey, and (4) complete another survey (on their own) 4-months after the baseline survey. Participants will complete a structured survey in the first meeting (baseline survey) with a member of the research team and then they will complete the follow-up surveys (1-month and 4-months after baseline) on their own.

Participants can request help to complete these surveys with the help of the research team (online using Zoom or face to face if needed). The moment that participants will access the IA intervention will depend on the group to be assigned by the research team (intervention or control group).

DETAILED DESCRIPTION:
Background Information Latinas continue to be affected disproportionally by HIV in the US.1 In 2017, Latinas accounted for 16% of new HIV diagnoses infection among women, a rate four-fold that of White women. To address this marked disparity, an innovative intervention - a filmed dramatized story (telenovela/soap opera) Infección de Amor (IA), or "Love Infection" - culturally tailored for US Latinas and delivered online is proposed in this study. IA is a four-episode HIV prevention telenovela co-created with Latinas and a community-based participatory and interdisciplinary. IA emphasizes the influence of romantic relationships in HIV infection and is available in Spanish and English. The development of IA incorporated the National Institute on Minority Health and Health Disparities (NIMHD) Framework, conceptualizing factors relevant to the understanding and promotion of minority health and understanding and reducing health disparities, to guide its content. Social cognitive theory, narrative engagement theory, and research on emotional responses are the mechanisms of action-guiding IA's delivery.

Participants A total of 66 Latinas ages 18-44 years who report sexual activity with a man in the last 6 months, have internet access from any device, and reside in NC.

Recruitment and screening will be led by a bilingual (English and Spanish) study personnel. Participants will be asked their preferred language at the time of recruitment. All study materials, including information and consent forms, questionnaires, and recruitment ads, will be translated and available in Spanish. Any direct interaction with non-English-speaking participants will be available in Spanish

Study procedures

The research team is bilingual and will be able to assist women if they have questions about the study. Study procedures will be conducted in English and/or Spanish according to participant's preference. A screening form to see if a person qualifies for the study that is available in Qualtrics will be used. If the person qualifies for the study, a first meeting to conduct the baseline survey will be arranged with the research team.

- Baseline survey. If potential participants meet the inclusion criteria, they will be asked to attend to a one hour-meeting with a member of the research team to sign the informed consent, complete a baseline survey and receive an orientation about the use of the telenovela website https://www.infecciondeamor.com/. After participants complete the survey, they will be randomized by a member of the research team to the intervention or control group. The research team member will explain the following activities they have to complete according to the group they will be assigned. If they are randomized to the control group, the orientation to the website will be delayed until they complete the 4-month post baseline survey. The survey will be available in Qualtrics and only the members of the research team will have access to the survey.

After completing the baseline survey, participants will be randomized to the intervention or control groups by a computer-generated randomization table, using blocking of participants to ensure a balance between groups. An envelope will contain the result of the randomization and the assessors will open this envelop in front of the participant after she finished the baseline survey. Each participants envelop will be assigned based on the ID number (e.g., 1, 2, 3)

- Intervention group: Latinas will view four IA intervention episodes, one per week. Participants will receive an email to their preferred email address with a password to access to the episode on the IA's website: https://www.infecciondeamor.com/ Each 10-minute episode can be watched more than once during the week and presents a situation with notable HIV risk and ways the characters avoided risk (e.g., condom use) or confronted consequences of poor practices (e.g., HIV infection).

After each episode, participants will complete a survey (on their own) on Qualtrics.

This post episode survey includes questions about the mechanisms of action of the telenovela (self-efficacy, narrative engagement, and emotional elicitation).

* Control group: A wait-listed control group of 33 Latinas will receive IA in the same manner as the intervention group after completing T3 data collection. During the waiting time, participants will be contacted on a monthly basis to encourage participation and refer to services if needed.
* Follow-up surveys. Participants will answer a (one-month after baseline) survey, and complete another survey (on their own) 4 months after baseline. Participants will complete these surveys (1-month and 4-months after baseline) on their own. Participants can request help to complete these surveys (online using zoom or face to face if needed).
* Infección de Amor website. The website provides: a) access to the four intervention episodes 24/7 from any location or type of device (e.g., cellphone, laptop) since is mobile optimized (all the episodes are password protected); b) questionnaires for data collection deployed via Qualtrics; c) a contact section; and d) a section with community resources, services, and referrals. Secure and private servers and communication channels such as OneDrive will be used to store and to exchange information.

A new episode of IA will be available each week. Women can watch an episode as many times as they want during the week, but they need to answer a post episode-viewing survey after viewing it the first time. Also, they will be able to pause or stop the episodes at any time if they need to take a break or stop watching for any reason. Women will be advised to watch the episodes alone. Prior episodes will remain available after a new episode is released. Participants will receive reminders about completion of the surveys using an automated notification system from Qualtrics. In addition, up to three reminders (e.g., phone, email) will be sent each week to participants who have not accessed an episode in a specific window period and completed the post episode survey or if the participant has not access to the website in one week. If a woman does not complete the episode in one week or does not access the website in one week, the research team will contact the participant to her preferred email or phone. The research team will discuss with her any impediments to her participation, how to watch the missed episode, and resume with the following episodes. Women will be able to pause or stop the episodes at any time if they need it. Prior episodes will remain available after a new episode is released if women would like to review them.

- Procedures for Minority Retention and Potential Challenges. The website will track if participants watched the whole episode. Each episode also contains information about HIV prevention at the end and a link to the technical support and referrals sections if needed. Other retention strategies will include: 1) updating contact information frequently; 2) requesting contact information of at least two friends or relatives; 3) contacting the woman by email or cell phone (permission to contact the participants will be requested in the informed consent); 4) providing compensation for their time, internet use, and transportation; and 5) automated notification system messages for special occasions (e.g., holidays). Attrition will be monitored in both conditions. Potential issues with Latinas and community centers, and if needed, establish a community advisory board of three Latinas of the same age as those participating in the study to ask for their advice.

Follow-up procedures Participants will have access to watch the intervention online individually 24/7 from their preferred location. They will be asked to watch the intervention in a comfortable and private place since some of the content (e.g., IPV, substance use) can be sensitive for them or other people (e.g., their children) if they allow them to watch. Participants will have a contact section on the online platform in case they have questions, they need referrals, or they want to talk about issues that may arise while they are watching the telenovela. If they are watching the telenovela and they experience stress or anxiety, they will be instructed to call a person from the team who will be available to listen to them and refer them to proper services if needed. The person from the team will notify the PI about the situation and how it should be managed. A protocol will be created by the research team to manage these situations. Latinas will be instructed that they can stop their participation at that moment and that this situation will not affect their ability to continue in the study.

Potential risks

The research team will treat Latinas with respect and will be sensitive if they express that they feel or voice embarrassment with the intervention content. The research team will explain to them that this will not affect their ability to continue in the study. If a potential breach of confidentiality occurs, which could be related with someone finding out that a participant is involved in the study or if a study member unintentionally disclosures confidential information about the participants. Efforts will be made to avoid these situations, by not revealing any information about participants to any people external to the research unless requested by authorities. Participants will be requested to keep their randomization to the groups (intervention or control) confidential. In addition, all the team members will have their Human subject training up to date and will receive a training to avoid situations that can lead to breach in confidentiality. .

Referrals El Futuro is a community center who provides mental health services to the Latino population. El Futuro will provide the space for the study related activities and will facilitate recruitment (flyers). In need of a referral, participants will be advised to call to this community center. A list of referrals to other community centers that provide culturally sensitive services in case they need other type of services (e.g., HIV test) will also be provided.

The Investigators will be responsible for ensuring that study protocols for maintaining confidentiality are followed. The PI will provide ongoing supervision and training to essential study staff at weekly meetings, which will also ensure continued compliance with data safety protocols.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified as a Latina
* Assigned female gender at birth
* Fluent in English or Spanish
* Between 18 and 44 years old
* Report sexual activity with a man in the last 6 months
* Have internet access from any device
* Reside in NC

Exclusion Criteria:

* Unwilling to be part of the study
* Do not read, speak, or understand Spanish or English
* Do not have access to internet
* HIV positive

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study includes female Latinas between 18 and 44 years old. Older women (>44 years old) and younger children/adolescents (<18) are excluded.
Enrollment: 58 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Villegas Rodriguez, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- El Futuro, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and continuing for 36 months following publication
Access Criteria: Borrower has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Background] Villegas N, Norris A, Cianelli R. Reducing disparities in HIV prevention: A telenovela for young Latina seasonal farmworkers in south Florida. CFAR pilot award. The Miami Center for AIDS Research (CFAR) at the University of Miami Miller School of Medicine (NIH grant number P30AI073961). 2017-2019.
- [Background] Larkey LK, Hecht ML, Miller K, Alatorre C. Hispanic cultural norms for health-seeking behaviors in the face of symptoms. Health Educ Behav. 2001 Feb;28(1):65-80. doi: 10.1177/109019810102800107. PMID 11213143
- [Background] Miller-Day M, Hecht ML. Narrative means to preventative ends: a narrative engagement framework for designing prevention interventions. Health Commun. 2013;28(7):657-70. doi: 10.1080/10410236.2012.762861. Epub 2013 Aug 27. PMID 23980613
- [Background] Dillard J, Peck E. Affect and persuasion: Emotional responses to public service announcements. Commun Res. 2000;27(4):461-495.
- [Background] North Carolina Department of Health and Human Services. 2018 North Carolina HIV surveillance report. HIV/STD/hepatitis surveillance unit division of public health North Carolina department of health and human services. https://epi.dph.ncdhhs.gov/cd/stds/figures/hiv18rpt_02042020.pdf. Updated 2019.
- [Background] Geter Fugerson A, Sutton MY, Hubbard McCree D. Social and Structural Determinants of HIV Treatment and Care Among Hispanic Women and Latinas Living with HIV Infection in the United States: A Qualitative Review: 2008-2018. Health Equity. 2019 Nov 4;3(1):581-587. doi: 10.1089/heq.2019.0039. eCollection 2019. PMID 31701083
- [Background] Hernandez AM, Zule WA, Karg RS, Browne FA, Wechsberg WM. Factors That Influence HIV Risk among Hispanic Female Immigrants and Their Implications for HIV Prevention Interventions. Int J Family Med. 2012;2012:876381. doi: 10.1155/2012/876381. Epub 2012 Feb 8. PMID 22518308
- [Background] Levison JH, Bogart LM, Khan IF, Mejia D, Amaro H, Alegria M, Safren S. "Where It Falls Apart": Barriers to Retention in HIV Care in Latino Immigrants and Migrants. AIDS Patient Care STDS. 2017 Sep;31(9):394-405. doi: 10.1089/apc.2017.0084. PMID 28891715
- [Background] Cianelli R, Ferrer L, McElmurry BJ. HIV prevention and low-income Chilean women: machismo, marianismo and HIV misconceptions. Cult Health Sex. 2008 Apr;10(3):297-306. doi: 10.1080/13691050701861439. PMID 18432428
- [Background] Villar-Loubet OM, Vamos S, Jones DL, Lopez E, Weiss SM. A Cultural Perspective on Sexual Health: HIV Positive and Negative Monolingual Hispanic Women in South Florida. Hisp Health Care Int. 2011 Jun 1;9(2):82-90. doi: 10.1891/1540-4153.9.2.82. PMID 24994949
- [Background] Cianelli R, Villegas N. Social Determinants of Health for HIV Among Hispanic Women. Hisp Health Care Int. 2016 Mar;14(1):4-9. doi: 10.1177/1540415316629672. No abstract available. PMID 27257185
- [Background] Sanchez M, Rojas P, Li T, Ravelo G, Cyrus E, Wang W, Kanamori M, Peragallo NP, De La Rosa MR. Evaluating a Culturally Tailored HIV Risk Reduction Intervention Among Latina Immigrants in the Farmworker Community. World Med Health Policy. 2016 Sep;8(3):245-262. doi: 10.1002/wmh3.193. Epub 2016 Sep 17. PMID 29034116
- [Background] Torrone EA, Wright J, Leone PA, Hightow-Weidman LB. Pregnancy and HIV infection in young women in North Carolina. Public Health Rep. 2010 Jan-Feb;125(1):96-102. doi: 10.1177/003335491012500113. PMID 20402201
- [Background] Paz K, Massey KP. Health Disparity among Latina Women: Comparison with Non-Latina Women. Clin Med Insights Womens Health. 2016 Jul 20;9(Suppl 1):71-4. doi: 10.4137/CMWH.S38488. eCollection 2016. PMID 27478393
- [Background] Garcia J, Perez-Brumer AG, Cabello R, Clark JL. "And Then Break the Cliche": Understanding and Addressing HIV Vulnerability Through Development of an HIV Prevention Telenovela with Men Who Have Sex with Men and Transwomen in Lima, Peru. Arch Sex Behav. 2018 Oct;47(7):1995-2005. doi: 10.1007/s10508-017-1119-x. Epub 2018 Feb 20. PMID 29464455
- [Background] Villegas N, Santisteban D, Cianelli R, Ferrer L, Ambrosia T, Peragallo N, Lara L. The development, feasibility and acceptability of an Internet-based STI-HIV prevention intervention for young Chilean women. Int Nurs Rev. 2014 Mar;61(1):55-63. doi: 10.1111/inr.12080. PMID 24512261
- [Background] Zou B, Jin B, Koch GG, Zhou H, Borst SE, Menon S, Shuster JJ. On model selections for repeated measurement data in clinical studies. Stat Med. 2015 May 10;34(10):1621-33. doi: 10.1002/sim.6414. Epub 2015 Jan 23. PMID 25645442
- [Result] Nabi R. Discrete emotions and persuasion. In: Dillard J, Pfau M, eds. The persuasion handbook: Developments in theory and practice. Thousand Oaks, CA: Sage; 2002:289-308.
- [Result] Nabi R. The persuasion handbook: Developments in theory and practice. In: Dillard J, Pfau M, eds. Thousand Oaks: Sage; 2002:289-308.
- [Result] Nabi RL. Emotional flow in persuasive health messages. Health Commun. 2015;30(2):114-24. doi: 10.1080/10410236.2014.974129. PMID 25470436
- [Result] Nabi RL. Laughing in the Face of Fear (of Disease Detection): Using Humor to Promote Cancer Self-Examination Behavior. Health Commun. 2016 Jul;31(7):873-83. doi: 10.1080/10410236.2014.1000479. Epub 2015 Dec 11. PMID 26652312
- [Result] Peragallo N, Deforge B, O'Campo P, Lee SM, Kim YJ, Cianelli R, Ferrer L. A randomized clinical trial of an HIV-risk-reduction intervention among low-income Latina women. Nurs Res. 2005 Mar-Apr;54(2):108-18. doi: 10.1097/00006199-200503000-00005. PMID 15778652
- [Result] Peragallo Montano N, Cianelli R, Villegas N, Gonzalez-Guarda R, Williams WO, de Tantillo L. Evaluating a Culturally Tailored HIV Risk Reduction Intervention Among Hispanic Women Delivered in a Real-World Setting by Community Agency Personnel. Am J Health Promot. 2019 May;33(4):566-575. doi: 10.1177/0890117118807716. Epub 2018 Oct 24. PMID 30354190
- [Result] Villegas N, Santisteban D, Cianelli R, Ferrer L, Ambrosia T, Peragallo N, Lara L. Pilot testing an internet-based STI and HIV prevention intervention with Chilean women. J Nurs Scholarsh. 2015 Mar;47(2):106-16. doi: 10.1111/jnu.12114. Epub 2014 Nov 19. PMID 25410132
- [Result] Cianelli R, Ferrer L, Norr KF, Miner S, Irarrazabal L, Bernales M, Peragallo N, Levy J, Norr JL, McElmurry B. Mano a Mano-Mujer: an effective HIV prevention intervention for Chilean women. Health Care Women Int. 2012;33(4):321-41. doi: 10.1080/07399332.2012.655388. PMID 22420675
- [Result] Sikkema KJ, Heckman TG, Kelly JA, Anderson ES, Winett RA, Solomon LJ, Wagstaff DA, Roffman RA, Perry MJ, Cargill V, Crumble DA, Fuqua RW, Norman AD, Mercer MB. HIV risk behaviors among women living in low-income, inner-city housing developments. Am J Public Health. 1996 Aug;86(8):1123-8. doi: 10.2105/ajph.86.8_pt_1.1123. PMID 8712272
- [Result] Heckman T, Kelly J, Sikkema K, et al. HIV risk characteristics of young adult, adult, and older adult women who live in inner-city housing developments: Implications for prevention. J Women's Health Gend Based Med. 1995;4(4):397-406.
- [Result] Garcia M, Harris AL. PrEP awareness and decision-making for Latino MSM in San Antonio, Texas. PLoS One. 2017 Sep 27;12(9):e0184014. doi: 10.1371/journal.pone.0184014. eCollection 2017. PMID 28953905
- [Result] Cianelli R, Villlegas N, De Oliveira G, Hires K, Gattamorta K, Ferrer L, Peragallo N. Predictors of HIV enacted stigma among Chilean women. J Clin Nurs. 2015 Sep;24(17-18):2392-401. doi: 10.1111/jocn.12792. Epub 2015 Feb 19. PMID 25693422
- [Result] Catania J. Dyadic sexual communication scale: Handbook of sexuality related measures. 1986.
- [Result] Catania JA, Kegeles SM, Coates TJ. Towards an understanding of risk behavior: an AIDS risk reduction model (ARRM). Health Educ Q. 1990 Spring;17(1):53-72. doi: 10.1177/109019819001700107. PMID 2318652
- [Result] Kelly JA, Murphy DA, Washington CD, Wilson TS, Koob JJ, Davis DR, Ledezma G, Davantes B. The effects of HIV/AIDS intervention groups for high-risk women in urban clinics. Am J Public Health. 1994 Dec;84(12):1918-22. doi: 10.2105/ajph.84.12.1918. PMID 7998630
- [Result] Straus MA, Douglas EM. A short form of the Revised Conflict Tactics Scales, and typologies for severity and mutuality. Violence Vict. 2004 Oct;19(5):507-20. doi: 10.1891/vivi.19.5.507.63686. PMID 15844722
- [Result] Radloff LS. The CES-D scale: A self-report depression scale for research in the general population. Appl Psychol Meas. 1977;1:385-401
- [Result] Card J, Solomon J, Berman J, eds. Tools for building culturally competent HIV prevention programs. New York: Springer Publishing Company; 2008.
- [Result] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Result] Lelutiu-Weinberger C, Golub SA. Enhancing PrEP Access for Black and Latino Men Who Have Sex With Men. J Acquir Immune Defic Syndr. 2016 Dec 15;73(5):547-555. doi: 10.1097/QAI.0000000000001140. PMID 27454250
- [Result] Bauermeister JA, Meanley S, Pingel E, Soler JH, Harper GW. PrEP awareness and perceived barriers among single young men who have sex with men. Curr HIV Res. 2013 Oct;11(7):520-7. doi: 10.2174/1570162x12666140129100411. PMID 24476355
- [Result] Walsh JL. Applying the Information-Motivation-Behavioral Skills Model to Understand PrEP Intentions and Use Among Men Who Have Sex with Men. AIDS Behav. 2019 Jul;23(7):1904-1916. doi: 10.1007/s10461-018-2371-3. PMID 30554396

RESULTS

PARTICIPANT FLOW:
Groups:
- Infeccion de Amor (Infectious Love): Participants will view four IA intervention episodes, one per week starting immediately after the baseline survey and orientation.
  Participants will receive an email to their preferred email address with a password to access the episode on the IA's website: https://www.infecciondeamor.com. Each 10-minute episode can be watched more than once during the week and presents a situation with notable HIV risk and ways the characters avoided risk (e.g., condom use) or confronted consequences of poor practices (e.g., HIV infection).
  Infeccion de Amor (Infectious Love): Infectious Love is a filmed dramatized story (telenovela/soap opera) Infección de Amor (IA), or "Infectious Love" - culturally tailored for US Latinas and delivered online. IA is a four-episode HIV prevention telenovela co-created with Latinas and a community-based participatory and interdisciplinary. Participants have one week window to watch the 10-minute episodes from their preferred device and location.
- Wait-listed: Participants will receive IA in the same manner as the intervention group.
  Participants will start watching the telenovela episodes 4 months after their baseline survey (after T3 survey). Participants will be informed at recruitment of this group condition and the study randomization. During the waiting time, participants will be called on a monthly basis to encourage participation and refer to services if needed.
  Infeccion de Amor (Infectious Love): Infectious Love is a filmed dramatized story (telenovela/soap opera) Infección de Amor (IA), or "Infectious Love" - culturally tailored for US Latinas and delivered online. IA is a four-episode HIV prevention telenovela co-created with Latinas and a community-based participatory and interdisciplinary. Participants have one week window to watch the 10-minute episodes from their preferred device and location.
Period: Overall Study
Arm/Group | Infeccion de Amor (Infectious Love) | Wait-listed
Started | 31 | 27
Completed Follow-Up 1 (Month 1) | 26 | 26
Completed Follow-Up 2 (Month 4) | 25 | 23
Completed | 25 | 23
Not Completed | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Infeccion de Amor (Infectious Love): Participants will view four IA intervention episodes, one per week starting immediately after the baseline survey and orientation.
  Participants will receive an email to their preferred email address with a password to access the episode on the IA's website: https://www.infecciondeamor.com. Each 10-minute episode can be watched more than once during the week and presents a situation with notable HIV risk and ways the characters avoided risk (e.g., condom use) or confronted consequences of poor practices (e.g., HIV infection).
- Total: Total of all reporting groups
Arm/Group | Infeccion de Amor (Infectious Love) | Wait-listed | Total
Number analyzed (Participants) | 31 | 27 | 58
Age, Continuous [Mean (Full Range); unit: years] | 33.26 [19 to 44] | 36.37 [20 to 44] | 34.71 [19 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 27 | 58
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 27 | 58
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 0 | 0 | 0
  White | 15 | 8 | 23
  More than one race | 13 | 15 | 28
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 27 | 58

OUTCOME MEASURES:

1. Primary Outcome: Mean Condom Use
Description: Condom use will be measured as the number of sexual episodes (oral, vaginal, or anal intercourse) in which condoms were used with a male partner in the last month.
Time Frame: baseline up to 4 months
Population: No Infeccion de Amor (Infectious Love) participants reported engaging in anal intercourse at baseline. Month 1 data are reported for those in this group who completed Follow-Up 1 assessment (immediately after intervention period completion). Wait-listed participants completed Month 1 assessment before watching intervention (4 months after baseline). Month 4 data are reported for each arm for those who completed the second Follow-Up.
Measure: Mean (Standard Deviation); unit: sexual episodes
Arm/Group | Infeccion de Amor (Infectious Love) | Wait-listed
Number analyzed (Participants) | 31 | 27
sexual episodes
  Baseline Oral | 0.50 (1.414) | 0.14 (0.535)
  Baseline Vaginal | 1.30 (2.562) | 0.52 (1.159)
  Baseline Anal Intercourse: number analyzed (Participants) | 0 | 27
  Baseline Anal Intercourse |  | 0 (0)
  Month 1 Oral: number analyzed (Participants) | 26 | 26
  Month 1 Oral | 0 (0) | 1.25 (2.927)
  Month 1 Vaginal: number analyzed (Participants) | 26 | 26
  Month 1 Vaginal | 1.50 (2.526) | 1.43 (2.243)
  Month 1 Anal Intercourse: number analyzed (Participants) | 26 | 26
  Month 1 Anal Intercourse | 0 (0) | 3.00 (0)
  Month 4 Oral: number analyzed (Participants) | 25 | 23
  Month 4 Oral | 0 (0) | 0.09 (0.302)
  Month 4 Vaginal: number analyzed (Participants) | 25 | 23
  Month 4 Vaginal | 2.25 (2.933) | 1.75 (3.768)
  Month 4 Anal Intercourse: number analyzed (Participants) | 25 | 23
  Month 4 Anal Intercourse | 0 (0) | 0 (0)

2. Primary Outcome: Number of Participants Who Report Change in PrEP Awareness
Description: Changes in PrEP awareness will be measured as the number of participants who self-report whether they know about PrEP medication (dichotomous question: yes/no)
Time Frame: Baseline up to 4 months
Population: Data are reported for all participants who reported this information.
Measure: Count of Participants; unit: Participants
Arm/Group | Infeccion de Amor (Infectious Love) | Wait-listed
Number analyzed (Participants) | 31 | 27
Participants
  Baseline-Yes | 7 | 2
  Baseline-No | 24 | 25
  Month 1-Yes: number analyzed (Participants) | 26 | 24
  Month 1-Yes | 20 | 1
  Month 1-No: number analyzed (Participants) | 26 | 24
  Month 1-No | 6 | 23
  Month 4-Yes: number analyzed (Participants) | 25 | 22
  Month 4-Yes | 16 | 2
  Month 4-No: number analyzed (Participants) | 25 | 22
  Month 4-No | 9 | 20

3. Primary Outcome: Number of Participants Who Report Change in PrEP Access
Description: Changes in PrEP access will be measured as the number of participants who report that they have access to PrEP (Possible responses: yes/no/don't know). Those participants who answered "Yes" to the PrEP awareness question were asked if they have access to PrEP.
Time Frame: baseline to 4 months
Population: The Overall Number of Participants Analyzed reflects the number of unique participants who provided data for any single timepoint. Participants were asked to provide a response at each timepoint although some participants did not provide a response each time they were asked. Data are reported for all responses received.
Measure: Count of Participants; unit: Participants
Arm/Group | Infeccion de Amor (Infectious Love) | Wait-listed
Number analyzed (Participants) | 22 | 4
Participants
  Baseline-Yes: number analyzed (Participants) | 7 | 2
  Baseline-Yes | 2 | 0
  Baseline-No: number analyzed (Participants) | 7 | 2
  Baseline-No | 4 | 1
  Baseline-Don't Know: number analyzed (Participants) | 7 | 2
  Baseline-Don't Know | 1 | 1
  Month 1-Yes: number analyzed (Participants) | 20 | 1
  Month 1-Yes | 2 | 0
  Month 1-No: number analyzed (Participants) | 20 | 1
  Month 1-No | 9 | 0
  Month 1--Don't Know: number analyzed (Participants) | 20 | 1
  Month 1--Don't Know | 9 | 1
  Month 4-Yes: number analyzed (Participants) | 16 | 2
  Month 4-Yes | 5 | 0
  Month 4-No: number analyzed (Participants) | 16 | 2
  Month 4-No | 4 | 1
  Month 4--Don't Know: number analyzed (Participants) | 16 | 2
  Month 4--Don't Know | 7 | 1

4. Primary Outcome: Number of Participants Who Report Changes in PrEP Use
Description: Changes in PrEP use will be measured as the number of participants who report that they have used PrEP (dichotomous question: yes/no). Those participants who answered "Yes" to the PrEP awareness question were asked about PrEP use.
Time Frame: baseline to 4 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Infeccion de Amor (Infectious Love) | Wait-listed
Number analyzed (Participants) | 22 | 4
Participants
  Baseline-Yes: number analyzed (Participants) | 7 | 2
  Baseline-Yes | 0 | 0
  Baseline-No: number analyzed (Participants) | 7 | 2
  Baseline-No | 7 | 2
  Month 1-Yes: number analyzed (Participants) | 20 | 1
  Month 1-Yes | 0 | 0
  Month 1-No: number analyzed (Participants) | 20 | 1
  Month 1-No | 20 | 1
  Month 4-Yes: number analyzed (Participants) | 16 | 2
  Month 4-Yes | 0 | 0
  Month 4-No: number analyzed (Participants) | 16 | 2
  Month 4-No | 16 | 2

5. Primary Outcome: Number of Participants Who Report Change in HIV Testing
Description: Changes in HIV testing will be measured as the number of participants who reported to have been tested for HIV in the last month.
Time Frame: baseline up to 4 months
Population: This question was only asked of participants who indicated having had a previous HIV test within 30 days before study entry.
Measure: Count of Participants; unit: Participants
Arm/Group | Infeccion de Amor (Infectious Love) | Wait-listed
Number analyzed (Participants) | 25 | 24
Participants
  Baseline-Yes | 6 | 3
  Baseline-No | 19 | 21
  Month 1-Yes: number analyzed (Participants) | 23 | 17
  Month 1-Yes | 3 | 2
  Month 1-No: number analyzed (Participants) | 23 | 17
  Month 1-No | 20 | 15
  Month 4-Yes: number analyzed (Participants) | 24 | 21
  Month 4-Yes | 3 | 4
  Month 4-No: number analyzed (Participants) | 24 | 21
  Month 4-No | 21 | 17

6. Primary Outcome: Mean Change in HIV Test Perception Score
Description: Changes in HIV testing perception will be measured with the willingness to take an HIV test measure scale. Scores range from 9-45. A higher score represents a higher willingness to take an HIV test.
Time Frame: baseline up to 4 months
Population: Participants were asked to complete the HIV Test Perception Score at each timepoint although some participants did not do so each time. Data are reported for all completed questionnaires.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Infeccion de Amor (Infectious Love) | Wait-listed
Number analyzed (Participants) | 31 | 27
score on a scale
  Baseline | 34.7 (3.83) | 35.7 (4.07)
  Month 1: number analyzed (Participants) | 26 | 21
  Month 1 | 34.6 (3.37) | 36.4 (3.25)
  Month 4: number analyzed (Participants) | 23 | 17
  Month 4 | 32.8 (5.82) | 36.1 (4.33)

7. Secondary Outcome: Mean Change in Substance Abuse Score
Description: Changes in substance abuse will be measured with the Substance abuse behaviors scale. Scores range from 0-35. A higher score represents a higher use of substances.
Time Frame: baseline up to 4 months
Population: Participants were asked to complete the Substance Abuse Behaviors Scale at each timepoint although some participants did not do so each time. Data are reported for all completed questionnaires.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Infeccion de Amor (Infectious Love) | Wait-listed
Number analyzed (Participants) | 31 | 27
score on a scale
  Baseline | 2.42 (3.65) | 0.78 (1.09)
  Month 1: number analyzed (Participants) | 25 | 24
  Month 1 | 2.32 (3.78) | 0.96 (1.30)
  Month 4: number analyzed (Participants) | 24 | 22
  Month 4 | 2.75 (3.67) | 1.23 (2.86)

8. Secondary Outcome: Mean Change in Intimate Partner Violence (IPV) Score
Description: Changes in IPV measured using the revised Conflict Tactics Scale to measure women's self-reported IPV in the previous 3 months (e.g., your partner insulted you). Scores range from 0-36 points. A higher score indicates higher levels of IPV.
Time Frame: baseline up to 4 months
Population: Participants were asked to complete the IPV at each timepoint although some participants did not do so each time. Data are reported for all completed questionnaires.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Infeccion de Amor (Infectious Love) | Wait-listed
Number analyzed (Participants) | 30 | 27
score on a scale
  Baseline | 2.27 (3.52) | 2.78 (4.57)
  Month 1: number analyzed (Participants) | 25 | 24
  Month 1 | 2.28 (5.56) | 1.96 (3.26)
  Month 4: number analyzed (Participants) | 24 | 20
  Month 4 | 1.79 (3.72) | 1.25 (1.83)

9. Secondary Outcome: Mean Change in Depression (PHQ-9) Score
Description: Changes in depression will be measured with the Patient Health Questionnaire (PHQ-9), a 9-item scale commonly used for depression screening in primary care and other health settings. Scores range from 0-27. A higher score indicates more depressive symptoms.
Time Frame: baseline up to 4 months
Population: Participants were asked to complete the PHQ-9 at each timepoint although some participants did not do so each time. Data are reported for all completed questionnaires.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Infeccion de Amor (Infectious Love) | Wait-listed
Number analyzed (Participants) | 31 | 27
score on a scale
  Baseline | 5.61 (3.97) | 4.04 (4.05)
  Month 1: number analyzed (Participants) | 26 | 24
  Month 1 | 5.65 (4.36) | 2.29 (3.34)
  Month 4: number analyzed (Participants) | 24 | 22
  Month 4 | 6.67 (6.40) | 2.36 (2.92)

10. Secondary Outcome: Number of Episodes Watched by Participants
Description: The online website will track if the 40-minutes of the intervention content is viewed and the number of participants who complete of all content will be calculated.
Time Frame: immediately after watching each 10-minute weekly episode for up to 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Infeccion de Amor (Infectious Love) | Wait-listed
Number analyzed (Participants) | 31 | 27
Participants
  Watched 0 Episodes | 2 | 18
  Watched 1 Episodes | 1 | 2
  Watched 2 Episodes | 2 | 0
  Watched 3 Episodes | 0 | 0
  Watched 4 Episodes | 26 | 7

11. Secondary Outcome: Number of Participants Who Are Retained Through All Study Timepoints
Description: The number of participants who completed all study assessment timepoints from start to finish.
Time Frame: baseline up to 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Infeccion de Amor (Infectious Love) | Wait-listed
Number analyzed (Participants) | 31 | 27
Participants | 26 | 23

12. Other Pre Specified Outcome: Mean Participant Acceptability With the Intervention Content Areas Based on a 5 Point Rating System
Description: Participants will be asked to rate each of the 9 content area using a 5-star rating system where 1 star is the lowest and 5 points is the highest rating. A mean of all ratings will be calculated. The closer the mean is to 5.0, the higher the satisfaction with the content areas. Scores range from 9-45. A higher score indicates a higher level of acceptability.
Time Frame: one-month after the baseline survey
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Change in Self-Efficacy for Condom Use
Description: Changes in Self-Efficacy will be measured using the HIV self-efficacy for condom use survey. Scores range from 7-28. A higher score indicates a higher level of self-efficacy for condom use.
Time Frame: baseline up to 1 month
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Change in Self-Efficacy for HIV Prevention
Description: Changes in Self-Efficacy will be measured using the HIV self-efficacy for HIV prevention behaviors survey. Scores range from 11-55. A higher score indicates a higher level of self-efficacy for HIV prevention behaviors.
Time Frame: baseline up to 1 month
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Change in Narrative Engagement
Description: Narrative engagement will be measured with the Perception of Narrative Performance Scale, which measures three dimensions of engagement: interest, realism, and identification. Scores range from 9-36. A higher score indicates a higher level of engagement.
Time Frame: baseline up to 1 month
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Change in Emotional Response
Description: Changes in emotional Response will be measured with the International Positive and Negative Affect Schedule Short Form (I-PANAS-SF). Scores range from 10-50. The higher scores indicate the tendency to experience a positive and negative mood.
Time Frame: baseline up to 1 month
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Feasibility of the Intervention
Description: Measured as the total number of sessions attended by the participants as a whole.
Time Frame: baseline up to 4 months
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Changes in HIV Knowledge
Description: Change in HIV knowledge will be measured via the HIV Knowledge Scale. The score ranges from 0-12 with a higher score indicating a higher level of HIV-related knowledge.
Time Frame: baseline up to 4 months
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Changes in STI (Sexually Transmitted Infections) Testing
Description: Changes in STI testing will be measured as the number of participants who reported to have been tested for a STI in the last month.
Time Frame: baseline up to 4 months
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Changes in Sexual Communication With Partner
Description: Change in sexual communication with partner will be measured via the Partner communication Scale (Catania et al., 1995). The score ranges from 0-10 with a higher score indicating a higher level of partner communication.
Time Frame: baseline up to 4 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the time participants signed informed consent through completion of last follow-up, approximately 4 months.
Arm/Group | Infeccion de Amor (Infectious Love) | Wait-listed
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/27
Other Adverse Events (participants affected / at risk) | 0/31 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-03): https://cdn.clinicaltrials.gov/large-docs/66/NCT05358366/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-16): https://cdn.clinicaltrials.gov/large-docs/66/NCT05358366/ICF_001.pdf